CLINICAL TRIAL: NCT06691425
Title: Stereotactic Body Radiation Therapy for Inoperable Non-metastasized Pancreatic Adenocarcinoma: a Randomized Phase II Study
Brief Title: Stereotactic Body Radiation Therapy for Inoperable Non-metastasized Pancreatic Adenocarcinoma
Acronym: TORPEDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Research Antwerp (Other)
Collaborators: Kom Op Tegen Kanker (Other); Naslund Medical AB (Unknown); Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO22014GZA
Record Dates: First submitted 2024-10-04; First posted 2024-11-15 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Non-metastasized Unresectable Pancreatic Carcinoma
Keywords: Pancreatic cancer; Randomized; stereotactic body radiation therapy; inoperable; non-metastasized
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Chemotherapy alone (Active Comparator): Patients in arm A will receive standard treatment, more specifically chemotherapy (mFOLFIRINOX or Gemcitabine/nab-paclitaxel) alone. After the 12 weeks of induction chemotherapy followed by randomization, these patients will receive further chemotherapy. A maximal total duration of 24 weeks of chemotherapy (including induction chemotherapy) will be administered for patients in arm A undergoing R0/R1 resection. Duration of chemotherapy for patients in arm A not undergoing R0/R1 resection is left at the discretion of the treating physician.
  Interventions: Drug: Chemotherapy
- Arm B: Chemotherapy with SBRT (Experimental): Patients in arm B will receive SBRT in addition to chemotherapy (mFOLFIRINOX or Gemcitabine/nab-paclitaxel). After the 12 weeks of induction chemotherapy followed by randomization, these patients will receive another month of chemotherapy. Fiducial markers are implanted (unless MR LINAC is used to deliver radiotharapy) prior to the administration of SBRT, which will start 14 days (+/- 1 week) after either the first day of the eighth cycle of mFOLFIRINOX or the fifteenth day of the fourth cycle of Gemcitabine/nab-paclitaxel. 5 fractions of 8 Gy will be delivered. SBRT is preferably followed by further chemotherapy. The maximal total duration of chemotherapy for these patients is 24 weeks.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: Chemotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT (5 x 8 Gy)
  Arms: Arm B: Chemotherapy with SBRT
Drug: Chemotherapy — Standard of care: mFOLFIRINOX or gemcitabine/nab-paclitaxel

SUMMARY:
This is a multicenter randomized phase II trial that aims to include 160 patients with a non-metastatic (localized), inoperable pancreatic tumor. The study will take place at multiple centers across Europe. The primary objective of the study is to demonstrate superiority in progression free survival (PFS) by adding stereotactic body radiation therapy (SBRT) to chemotherapy for patients with an inoperable non-metastasized pancreatic tumor. SBRT is a radiotherapy technique (i.e. destroying cancer cells by means of ionizing irradiation) in which tumors can be irradiated with a high radiation dose. Surrounding healthy tissue is thus spared to the maximum extent. The primary endpoint of the TORPEDO study is 2-year PFS defined as the percentage of patients who are free of disease progression at 110 weeks after the date when the patients were drawn into 2 treatment groups (i.e. randomization). Secondary outcomes are, among others, quality of life, acute and late toxicity (i.e. adverse events), metastasis-free survival, local progression-free survival, overall survival, subsequent resectability, R0 resection and surgical morbidity.

During the study, patients without disease progression after 3 months of induction chemotherapy will be randomized 1:1 to either treatment with chemotherapy or treatment with a combination of chemotherapy and SBRT (5 x 8 Gy). After randomization, ten-weekly follow-up visits will occur during two years to evaluate the quality of life, general blood parameters and general health condition of the patient. Moreover, toxicity will be evaluated as well as efficiency and safety of the treatment (e.g. by means of imaging). At any time during this follow-up period, imaging (CT scan, MRI scan) will be used to determine whether surgery can still be performed to improve patient survival.

DETAILED DESCRIPTION:
The occurrence of pancreatic cancer is increasing in Belgium. Although this type of cancer is severe, there are only a limited number of treatment options. The preferred treatment is usually surgery. However, this is only possible in certain circumstances. If surgery is not possible, chemotherapy is administered to improve survival. A combination of chemotherapy and SBRT followed by surgery if possible has already been used in some studies and will be investigated in a larger number of subjects with the TORPEDO study.

A patient needs to sign an informed consent form before participating in the TORPEDO study. Participation in the TORPEDO study consists of the following phases: screening, induction chemotherapy, restaging and randomization, treatment and a follow-up phase (during which resectability is multidisciplinary evaluated at any time).

During the screening phase, eligibility of the patient to participate in the study will be assessed. Demographics data, information regarding medical history, prior medications and adverse events will be recorded. Moreover, a clinical assessment, blood tests to assess general blood parameters, a CT chest/abdomen and MRI pancreas will be performed. Eligible patients (according to the inclusion criteria and exclusion criteria) will receive induction chemotherapy (standard of care) during 12 weeks. Either 6 cycles of mFOLFIRINOX or 3 cycles of gemcitabine / nab-paclitaxel will be administered. If at the end of 12 weeks of induction chemotherapy (restaging), CT chest/abdomen and MRI pancreas do not show extrapancreatic disease, in absence of massive gastric or intestinal invasion and if there is no known presence of an active ulcer, subjects will be randomized 1:1 to either treatment with chemotherapy (arm A) or treatment with a combination of chemotherapy and SBRT (5 x 8 Gy) (arm B).

Participants in arm A will be further treated with chemotherapy. Participants in arm B will be treated with an additional 4 weeks of chemotherapy (either 2 cycles of mFOLFIRINOX or 1 cycle of gemcitabine/nab-paclitaxel) before they proceed to SBRT (5 fractions of 8 Gy), preferably followed by further chemotherapy. A maximal total duration of 24 weeks of chemotherapy (including induction chemotherapy) will be administered for all patients in arm B (SBRT-arm) and for patients in arm A undergoing R0/R1 resection. Duration of chemotherapy for patients in arm A not undergoing R0/R1 resection is left at the discretion of the treating physician.

The follow-up phase consists of ten-weekly follow-up visits during 110 weeks (+/- 1 week). These follow-up visits consist of a clinical assessment, CT chest/abdomen imaging (and MRI pancreas during the first follow-up visit), blood sampling, elicitation of AE's and assessment of the subject's quality of life through questionnaires. After these 110 weeks, patients will be followed by standard of care, six monthly during the following 3 years. After five years, patients will be followed on a yearly basis (standard of care). Follow-up data (survival status) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be over 18 years of age.
* Participant is able and willing to provide written informed consent which includes compliance with and ability to undergo all study procedures and attend the scheduled follow-up visits per protocol.
* Either locally advanced or borderline resectable pancreatic adenocarcinoma, as confirmed by diagnostic images (CT, MRI or PET-CT scan) and based on vessel involvement according to the NCCN guidelines. Only borderline resectable pancreatic cancer (BRPC) patients who are medically unfit for surgery or refusing surgery can be included.
* Adequate organ function determined by the following laboratory values:

  * Adequate bone marrow function: absolute neutrophil count ≥1500/mm^3, platelet count ≥100000/mm^3 and hemoglobin ≥9 g/dl
  * Adequate renal function: Creatinine ≤1.5 x upper normal limit of normal (ULN) or estimated eGFR more than 45 ml/min
  * Adequate liver function: total bilirubin ≤1.5 ULN (after adequate biliairy stenting with metal stent) and alanine aminotransferase (ALT) ≤5x ULN
* An Eastern Cooperative Oncology Group (ECOG) performance status grade of 0-2.
* A life expectancy ≥3 months
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

  * Is not a woman of child bearing potential or
  * A woman of child bearing potential must have a negative serum pregnancy test at screening and must use a very effective method of birth control.

Exclusion Criteria:

* Extrapancreatic metastatic disease as defined on diagnostic imaging (CT, MRI or PET-CT scan) or laparoscopy, including distal nodal involvement beyond the peripancreatic tissues and/or distant metastases.
* Massive gastric or intestinal invasion as assessed on imaging and/or endoscopy. Direct invasion of the duodenal mucosa as visible on endoscopic ultrasound (EUS).
* Prior radiation therapy that could hamper adequate dose delivery
* Contraindication to magnetic resonance imaging (MRI)
* Diagnosis of another malignancy within 2 years prior to randomization, except non-melanoma skin cancer, non-invasive bladder cancer, carcinoma in situ of the cervix or non-metastatic prostate cancer. Patients with a history of other malignancies are eligible if they have been continuously disease-free for at least 2 years after definitive primary treatment.
* Any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject.
* Patient already included in another clinical trial that would interfere with the TORPEDO clinical trial, as assessed by the Investigator.
* Known presence of an active ulcer (i.e. detected during standard of care diagnostic assessments)

Additional exclusion criteria after restaging (i.e. within 1 week after 3 months of induction chemotherapy) and prior to randomization:

* Extrapancreatic metastatic disease as defined on diagnostic imaging, including distal nodal involvement beyond the peripancreatic tissues and/or distant metastases
* Massive gastric or intestinal invasion as assessed on imaging and/or endoscopy. Direct invasion of the duodenal mucosa as visible on EUS.
* Known presence of an active ulcer (i.e. detected during standard of care diagnostic assessments)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | From randomization until 110 weeks (+/- 1 week) after the date of randomization, assessed up to 110 weeks (+/- 1 week).
  2-year progression-free survival (PFS): defined as the percentage of patients who are free of disease progression at 110 weeks (+/- 1 week) after the date of randomization.
  Events considered as progression are:
  * Disease progression per RECIST 1.1 with the exception of cases determined as pseudoprogression at the first response assessment (i.e. at 10w +/- 1w after randomization).
  * Discovery of hepatic or peritoneal carcinomatosis during surgical exploration
  * Recurrent disease following R0/R1 resection
  * Death due to any cause

SECONDARY OUTCOMES:
Metastasis-free survival (MFS) | Measured from the date of randomization to time of distant metastasis, assessed up to 110 weeks (+/- 1 week)
  Survival without metastases
Local progression-free survival (LPFS) | Measured from the date of randomization to locoregional progression, assessed up to 110 weeks (+/- 1 week).
  Locoregional progression is defined as any progressive or recurrent pancreatic tumor at the original tumor location or the N1-2 lymph node areas (with the only exception of cases determined as pseudoprogression at the first restaging post SBRT).
Overall survival (OS) | Measured from the date of randomization to the date of death or last known follow-up date, assessed up to 6 years
  Overall survival
R0 resection rate | Measured at the moment surgery took place (if surgery took place)
  R0 resection rate is measured as the percentage of patients undergoing R0 resection. R0-resection is defined as a tumor-free margin of at least 1mm from the resection margins, with the exception for the anterior resection margin for which R0-resection is defined as the absence of tumor cells in the inked surface of the resection specimen.
Acute and late toxicity | From signing ICF until 110 weeks (+/- 1 week) after randomization, assessed up to approximately 2.5 years
  The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 will be used to classify and grade the intensity of adverse events (AEs) occurring until disease progression. Acute AEs are those occurring within 90 days after starting chemotherapy. Late AEs are those occurring more than 90 days after starting chemotherapy.
Subsequent resectability | At any time during follow-up (i.e. at any time during 110 weeks (+/- 1 week) after randomization)
  Resectability is determined after review of mp-MRI and CT scans and multidisciplinary discussion.
Surgical morbidity | Measured from randomization on until 110 weeks (+/- 1 week) after randomization
  On one hand, this includes rates of attempted resection, excluding "open and close" operations.
  On the other hand surgical complications: length of stay, death within 30 days, frequency and severity of adverse events at 30 and 90 days post surgery as defined according to the Clavien-Dindo classification and definitions of post pancreatic surgery complications (pancreatic fistula, delayed gastric emptying and bleeding) by the International Study group on Pancreatic Surgery.
Correlation between doses to organs at risk (OARs) and gastrointestinal toxicity | Only applicable in case of arm B: From simulation until 110 weeks (+/- 1 week) after randomization, assessed up to 110 weeks (+/- 1 week)
  Correlation between the doses to stomach, duodenum, small bowel and large bowel structures (maximal doses and dose constraints) and the rate of > G2 gastrointestinal toxicity as assessed per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be evaluated.
Correlation between planning target volume (PTV) coverage and delivered dose with local control, PFS and OS | Only applicable in case of arm B: From simulation until the end of follow-up, assessed up to 6 years.
  Correlation between PTV coverage and dose with local control, progression free survival (PFS) and overall survival (OS).
Quality of life measurement by EORTC QLQ-C30 questionnaire (specific functional dimensions / symptom items / single items) | From the start of induction chemotherapy until 110 weeks (+/- 1 week) after randomization, i.e. at following points: start induction chemotherapy, restaging, first and last SBRT fraction (arm B only), every 10-weekly follow-up visit.
  Mean changes in EORTC-QLQ-C30 scale scores regarding specific functional dimensions / symptom items / single items over time will be compared, both for change from baseline and absolute scores. The scale ranges from 1 up to 4 with a higher score indicating a worse outcome.
Quality of life measurement by EORTC QLQ-C30 questionnaire (overall health/overall quality of life) | From the start of induction chemotherapy until 110 weeks (+/- 1 week) after randomization, i.e. at following points: start induction chemotherapy, restaging, first and last SBRT fraction (arm B only), every 10-weekly follow-up visit.
  Mean changes in EORTC-QLQ-C30 scale scores regarding overall health / overall quality of life over time will be compared, both for change from baseline and absolute scores. The scale ranges from 1 up to 7 with a higher score representing a better outcome.
Quality of life measurement by EORTC QLQ-PAN26 questionnaire | From the start of induction chemotherapy until 110 weeks (+/- 1 week) after randomization, i.e. at following points: start induction chemotherapy, restaging, first and last SBRT fraction (arm B only), every 10-weekly follow-up visit.
  Mean changes in EORTC QLQ-PAN26 scale scores regarding disease symptoms/treatment side-effects/emotional issues specific to pancreatic cancer over time will be compared, both for change from baseline and absolute scores. The scale ranges from 1 up to 4 with a higher score indicating a worse outcome.
Objective response rate (ORR) assessed on imaging (multiparametric MRI (mp-MRI) and computed tomography (CT)) | Measured from enrollment in the study until 110 weeks (+/- 1 week) after randomization (more specifically measured at following timepoints: restaging, every ten-weekly follow-up visit).
  The objective response rate will be measured as the percentage of patients with a partial or complete response to treatment according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (9):
- Belgium (9):
  - UZA, Edegem, Antwerpen
  - ZAS Augustinus, Wilrijk, Antwerp
  - AZ Klina, Brasschaat
  - AZ Sint-Jan, Bruges
  - ZOL, Genk
  - Jessa ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout

REFERENCES:
- [Derived] Stas D, Vandamme T, Roeyen G, Reynders D, Demey W, Stellamans K, Bussels B, Hutsebaut I, Maurissen I, Bouchart C, Berbee M, Lallemand F, Poels H, Thomas M, Cuyle PJ, Bulens P, Verboven K, Martens M, Weytjens R, Joye I. Stereotactic body radiation therapy for inoperable non-metastasized pancreatic adenocarcinoma: a randomised phase II study (TORPEDO). BMC Cancer. 2025 Oct 30;25(1):1671. doi: 10.1186/s12885-025-15041-8. PMID 41168707